CLINICAL TRIAL: NCT05477303
Title: Artificial Intelligence to Evaluate Postoperative Pain Based on Facial Expression Recognition and Analgesia Nociception Index
Brief Title: Artificial Intelligence to Evaluate Postoperative Pain Based on Facial Expression
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Park InSun, Clinical instructor, Seoul National University Bundang Hospital
Other Study IDs: B-2205-757-304
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Artificial Intelligence; Facial Expression; Analgesia; Pain, Postoperative
MeSH Terms: conditions — Facial Expression; Agnosia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: taking a picture of a painful facial expression — Immediately after surgery, the patient's facial expression and the NRS score and ANI score reported by the patient are checked together.

SUMMARY:
Patients' subjective complaints about pain intensity are difficult to objectively evaluate, and may lead to inadequate pain management, especially in patients with communication difficulties.

DETAILED DESCRIPTION:
Analgesia nociception index (ANI 0-100) and patient-reported numeric rating scale (NRS 0-10) were trained on a convolutional neural network (CNN) model by linking the patients' facial expression with the score. By applying the predicted pain score by the AI model to evaluate pain, it is intended to measure the intensity of pain in an automatic, fast, and objective way for appropriate pain management.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19-75 years who were scheduled for elective laparoscopic abdominal surgery under general anesthesia
* American Society of Anesthesiology (ASA) class I-II

Exclusion Criteria:

* Patients who have difficulty in communicating and reporting pain
* Underlying diseases: liver, kidney, brain
* Patients with BMI greater than 30 and less than 18.5
* Alcohol or drug dependent patients
* Patients with severe or acute respiratory failure
* Opioid, NSAID allergy
* Patients who are scheduled to be admitted to the intensive care unit after surgery
* Patients who undergo cooperative surgery

Ages: 19 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were scheduled for elective laparoscopic abdominal surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-04-20 (Estimated); Study Completion 2026-05-09 (Estimated)

PRIMARY OUTCOMES:
Facial expression | immediately preoperative, postoperative time
  Painful facial expression
analgesia nociception index | immediately preoperative, postoperative time
  ANI score
numeric rating scale | immediately preoperative, postoperative time
  pain score

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyunggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park I, Park JH, Yoon J, Na HS, Oh AY, Ryu J, Koo BW. Machine learning model of facial expression outperforms models using analgesia nociception index and vital signs to predict postoperative pain intensity: a pilot study. Korean J Anesthesiol. 2024 Apr;77(2):195-204. doi: 10.4097/kja.23583. Epub 2024 Jan 5. PMID 38176698
- [Derived] Park I, Park JH, Yoon J, Song IA, Na HS, Ryu JH, Oh AY. Artificial intelligence model predicting postoperative pain using facial expressions: a pilot study. J Clin Monit Comput. 2024 Apr;38(2):261-270. doi: 10.1007/s10877-023-01100-7. Epub 2023 Dec 27. PMID 38150126